CLINICAL TRIAL: NCT03518996
Title: Non-Invasive Brain Stimulation and Delirium
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Gen Shinozaki (Other)
Responsible Party: Sponsor-Investigator, Gen Shinozaki, Associate Professor of Psychiatry, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201803846
Record Dates: First submitted 2018-04-17; First posted 2018-05-08 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Mental Disorders; Delirium
MeSH Terms: conditions — Mental Disorders; Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TMS/tACS (Experimental): Subjects will receive 5 days of 3x daily rTMS (intermittent theta burst stimulation) or tACS (transcranial alternating current stimulation) targeted over the cerebellum.
  Interventions: Device: rTMS/iTBS/tACS
- Sham TMS/tACS (Sham Comparator): Subjects will receive 5 days of 3x daily sham stimulation of the cerebellum.
  Interventions: Device: Sham TMS/tACS

INTERVENTIONS:
Device: rTMS/iTBS/tACS — Subjects with delirium and matched-controls will be receive theta frequency stimulation of the cerebellum. We will target the cerebellar vermis.
  Arms: TMS/tACS
Device: Sham TMS/tACS — Subjects with delirium and matched-controls will be receive sham stimulation of the cerebellum. We will target the cerebellar vermis.
  Other Names: Sham stimulation
  Arms: Sham TMS/tACS

SUMMARY:
The purpose of this study is to examine whether non-invasive brain stimulation can be used to improve cognitive deficits in patients with delirium.

DETAILED DESCRIPTION:
Data from subject's EPIC medical record will be abstracted for use in research analysis - the following elements will be reviewed: Information regarding diagnosis, age, gender, ethnicity/race, medication they are receiving as well as their past medical history, and DOSS score. The study team member will also discuss patient's mental status with their treating clinician before approaching him/her. The treating clinician will be consulted and must agree that it is appropriate for the delirious patient to be approached for enrollment. Beforehand, a clinician on the research team (Dr. Gen Shinozaki) will evaluate the subjects ability to sign consent, and thus, whether they can be approached for enrollment.

When subject is identified, consent team will approach to obtain consent (and assent when applicable), email address and research demographic information. If consented, subject undergo a short CAM-ICU assessment of delirium indication - the CAM-ICU is a delirium screening tool and is not done for screening individuals out of the study, a cognitive function evaluation (MoCA), Clinical Dementia Rating (CDR), and a longer delirium evaluation (DRS-R-98) conducted by a study team member.

Next, study personnel will obtain buccal swab samples and will assist with saliva samples. Trained medical staff will perform the blood draw for the blood collection sample, approximately 5-10 mL of blood per sample will be collected. If consented, subject will be asked to wear non-invasive EEG device (with two standard, clinical leads) on their head at the time of initial evaluation and up to two times daily during their hospital stay. What subjects will be asked to do/what happens in the study (in sequential order) if they meet inclusion criteria and consent, they will be asked to wear non-invasive EEG device (with two standard, clinical leads) on their head with EEG monitor capability up to three times daily while they are in the hospital.

One session of non-invasive brain stimulation will be administered. Study personnel will again obtain buccal swab samples and will assist with saliva samples. Trained research team members will perform the blood draw for the blood collection sample, approximately 5-10 mL of blood per sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis consistent with enrollment (positive for delirium)

Exclusion Criteria:

* History of recurrent seizures or epilepsy
* Any other neurological or psychiatric diagnosis outside the diagnosis for which the participant is enrolled.
* Active substance use disorder in the past 6 months other than tobacco use disorder.
* Pacemaker
* Coronary Stent
* Defibrillator
* Neurostimulation
* Claustrophobia
* Uncontrolled high blood pressure
* Atrial fibrillation
* Significant heart disease
* Hemodynamic instability
* Kidney disease
* Pregnant, trying to become pregnant, or breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in brain rhythms | During the 1 week of treatment, with follow up 1 week
  Change from baseline EEG activity in participants receiving stimulation

SECONDARY OUTCOMES:
Delirium Observation Screening (DOS) Scale | During the 1 week of treatment, with follow up 1 week
  Change between pre- and post-intervention DOS assessment (disease-specific symptom rating scale); The Delirium Observation Screening (DOS) Scale is a screen designed to allow faster, easier identification of delirium. The DOS is a 13-point screen for delirium (range 0-9). Higher values represent a worse outcome (scores greater than or equal to 3 are usually considered positive delirium screens).
Delirium Rating Scale-R-98 (DRS) | During the 1 week of treatment, with follow up 1 week
  Change between pre- and post-intervention DRS assessment (disease-specific symptom rating scale); The Delirium Rating-Scale-Revised-98 (DRS-R-98) is an instrument which has provision for assessment of broad range of symptoms of delirium. The instrument has a total range of 0-20.
  The severity ratings range from 0 (no impairment) to 3 (severe impairment) and a severity score > 15 or a total score of > 18 is indicative of delirium; higher scores indicate higher severity of delirium.
Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) | During the 1 week of treatment, with follow up 1 week
  Change between pre- and post-intervention CAM-ICU assessment; Confusion Assessment Method for the ICU (CAM-ICU). CAM-ICU is a valid and reliable delirium assessment tool recommended by the Society of Critical Care Medicine (SCCM) in its 2013 Pain, Agitation, and Delirium (PAD) guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Gen Shinozaki, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Marcantonio ER. Postoperative delirium: a 76-year-old woman with delirium following surgery. JAMA. 2012 Jul 4;308(1):73-81. doi: 10.1001/jama.2012.6857. PMID 22669559
- [Background] Flinn DR, Diehl KM, Seyfried LS, Malani PN. Prevention, diagnosis, and management of postoperative delirium in older adults. J Am Coll Surg. 2009 Aug;209(2):261-8; quiz 294. doi: 10.1016/j.jamcollsurg.2009.03.008. Epub 2009 May 1. No abstract available. PMID 19632604
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702
- [Background] Numata S, Ye T, Hyde TM, Guitart-Navarro X, Tao R, Wininger M, Colantuoni C, Weinberger DR, Kleinman JE, Lipska BK. DNA methylation signatures in development and aging of the human prefrontal cortex. Am J Hum Genet. 2012 Feb 10;90(2):260-72. doi: 10.1016/j.ajhg.2011.12.020. Epub 2012 Feb 2. PMID 22305529
- [Background] Sen P, Shah PP, Nativio R, Berger SL. Epigenetic Mechanisms of Longevity and Aging. Cell. 2016 Aug 11;166(4):822-839. doi: 10.1016/j.cell.2016.07.050. PMID 27518561
- [Background] Tsai PC, Spector TD, Bell JT. Using epigenome-wide association scans of DNA methylation in age-related complex human traits. Epigenomics. 2012 Oct;4(5):511-26. doi: 10.2217/epi.12.45. PMID 23130833
- [Background] Christensen BC, Houseman EA, Marsit CJ, Zheng S, Wrensch MR, Wiemels JL, Nelson HH, Karagas MR, Padbury JF, Bueno R, Sugarbaker DJ, Yeh RF, Wiencke JK, Kelsey KT. Aging and environmental exposures alter tissue-specific DNA methylation dependent upon CpG island context. PLoS Genet. 2009 Aug;5(8):e1000602. doi: 10.1371/journal.pgen.1000602. Epub 2009 Aug 14. PMID 19680444
- [Background] Day K, Waite LL, Thalacker-Mercer A, West A, Bamman MM, Brooks JD, Myers RM, Absher D. Differential DNA methylation with age displays both common and dynamic features across human tissues that are influenced by CpG landscape. Genome Biol. 2013;14(9):R102. doi: 10.1186/gb-2013-14-9-r102. PMID 24034465
- [Background] Barrientos RM, Higgins EA, Biedenkapp JC, Sprunger DB, Wright-Hardesty KJ, Watkins LR, Rudy JW, Maier SF. Peripheral infection and aging interact to impair hippocampal memory consolidation. Neurobiol Aging. 2006 May;27(5):723-32. doi: 10.1016/j.neurobiolaging.2005.03.010. PMID 15893410